CLINICAL TRIAL: NCT06994975
Title: CHinese ischEmic Stroke Beyond 4.5 Hours With TeNecteplase Under Optimized Non-Contrast CT Selection
Acronym: CHESTNUT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xin Cheng, Professor and Vice Chair, Department of Neurology, Huashan Hospital, Fudan University, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-720
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, blinded-endpoint, randomized, controlled, phase 3 trial
Who Masked: Outcomes Assessor
Masking Description: Blinded-endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.25mg/kg TNK group (Experimental)
  Interventions: Drug: 0.25mg/kg TNK
- Standard medical treatment (Placebo Comparator)
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Drug: 0.25mg/kg TNK — Patients in the tenecteplase group were administered a 0.25mg/kg dose as a bolus over 5-10 seconds, followed by a 2 mL saline flush.
  Arms: 0.25mg/kg TNK group
Drug: Standard medical treatment — Patients in the standard medical treatment group will receive the standard treatment selected by local doctors, including antithrombotic agents, lipid-lowering agents, antihypertensive drugs, and hypoglycemic agents. Patients would be ineligible if bridging endovascular treatment is planned at the time of randomization.
  Arms: Standard medical treatment

SUMMARY:
The CHESTNUT trial is a multicenter, open-label, blinded-endpoint, randomized, controlled, phase 3 trial. The primary objective of this study is to explore the efficacy and safety of the dose of 0.25 mg/kg tenecteplase (TNK) in Chinese acute ischemic stroke (AIS) patients without substantial infarction on non-contrast computed tomography (NCCT) in an extended time window.

DETAILED DESCRIPTION:
CHinese ischEmic Stroke beyond 4.5 Hours with TeNecteplase Under optimized Non-Contrast CT selection (CHESTNUT) is a multicenter, open-label, blinded-endpoint, randomized, controlled, phase 3 study. Patients with acute strokes who are unable to undergo endovascular thrombectomy and exhibit no substantial infarction lesion on non-contrast computed tomography (less than 50 mL according to the automated NCCT post-processing model and no visible hypodensity in more than 1/3 of the middle cerebral artery [MCA] territory) are randomly assigned in a 1:1 ratio to receive either 0.25 mg/kg TNK or standard medical treatment. The efficacy and safety of 0.25 mg/kg TNK are assessed through clinical prognosis at 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected acute ischemic stroke of anterior cerebral circulation.
2. Last known well time >4.5 hours.
3. Age ≥18 years old.
4. Baseline NIHSS (National Institutes of Health Stroke Scale) score >5.
5. Premorbid modified Rankin Scale (mRS) ≤1.
6. Imaging criteria: Automated infarct segmentation by NCCT post-processing model indicates infarct core volume <50 mL with no visible hypodensity in >1/3 of the MCA territory.
7. Informed consent signed by the patient or the patient's legally authorized representative.

Exclusion Criteria:

1. Obvious hypodensity on NCCT deemed related with the current stroke event, with no expected benefit from thrombolysis as assessed by the investigators
2. Endovascular thrombectomy (EVT) planned at the time of randomization
3. Allergy to the test drug and its ingredients
4. Rapidly improving symptoms at the discretion of the investigator
5. Any sign of an acute intracranial hemorrhage or subarachnoid hemorrhage identified on baseline NCCT
6. History of any intracranial hemorrhage
7. History of ischemic stroke or major head trauma within the last 3 months
8. History of intracranial/intraspinal surgery during the last 3 months
9. Gastrointestinal malignancy or gastrointestinal bleeding within 21 days
10. Known bleeding diatheses; platelets count < 100000/mm3, international normalized ratio > 1.7, prothrombin time > 15 s, or activated partial thromboplastin clotting time > 40 s
11. Treatment with a full dosage of low-molecular weighted heparin in the last 24 hours
12. Treatment with direct thrombin inhibitors or direct factor Xa inhibitors within the previous 48 hours unless the laboratory test of coagulation function is normal
13. Initial systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg
14. Initial glucose levels <2.8 or 22.22 mmol/L
15. Known or suspected aortic arch dissection

In addition to:

1. Clinical presentation or imaging profile consistent with Moyamoya disease/syndrome.
2. Pregnancy or breastfeeding.
3. Recent participation in another investigational drug or device study or registry in the past 30 days before enrollment.
4. Any terminal illness such that the patient would not be expected to survive more than three months.
5. Other conditions in which investigators believe that participating in this study may be harmful to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Excellent Functional Outcome (mRS 0-1) at 90±7 Days | at 90±7 days
  The primary outcome is the proportion of participants achieving excellent functional outcome (free of disability, defined as a modified Rankin Scale [mRS] score of 0-1) at 90±7 days.

SECONDARY OUTCOMES:
Infarct Growth Volume at 3-5 Days Compared to Baseline Core | at 3-5 days
  The secondary radiological efficacy outcome is infarct growth, defined as the difference in volume between the infarct volume measured by diffusion-weighted imaging (DWI) or non-contrast head CT at 3-5 days and the baseline core infarct volume.
Proportion of Participants Achieving Good Functional Outcome (mRS 0-2) at 90±7 Days | at 90±7 days
  The secondary clinical efficacy outcome is the proportion of participants achieving good functional outcome (functional independence, defined as a modified Rankin Scale [mRS] score of 0-2) at 90±7 days.
Distribution of Modified Rankin Scale Scores at 90±7 Days | at 90±7 days
  The secondary clinical efficacy outcome is the distribution of modified Rankin Scale (mRS) scores from 0 (no symptoms) to 6 (death) at 90±7 days post-treatment.
Proportion of Participants with Significant Neurological Improvement within 24-48 Hours | within 24-48 hours
  The secondary clinical efficacy outcome is the proportion of participants achieving significant neurological improvement within 24-48 hours, defined as a reduction in National Institutes of Health Stroke Scale (NIHSS) score by more than 8 points or an NIHSS score of 0-1.
Change in NIHSS Score at 24-48 Hours | at 24-48 hours
  The secondary clinical efficacy outcome is the change in National Institutes of Health Stroke Scale (NIHSS) score as a continuous variable at 24-48 hours post-treatment.
Incidence of Symptomatic Intracranial Hemorrhage within 24-48 Hours | within 24-48 hours
  The secondary radiological safety outcome is the incidence of symptomatic intracranial hemorrhage within 24-48 hours post-treatment, defined according to the European Cooperative Acute Stroke Study III (ECASS III) criteria.
Incidence of Any Intracranial Hemorrhage within 24-48 Hours Post Treatment | at 24-48 hours
  The secondary radiological safety outcome is the incidence of any intracranial hemorrhage within 24-48 hours post-treatment, as determined by computed tomography [CT].
Incidence of PH2 within 24-48 Hours Post Treatment | at 24-48 hours
  The secondary radiological safety outcome is the incidence of type 2 parenchymal hematoma (PH2) within 24-48 hours post-treatment, as determined by computed tomography [CT].
Incidence of All-Cause Mortality within 90 Days | within 90 days
  The secondary clinical safety outcome is the incidence of all-cause mortality within 90 days post-treatment.
Proportion of Participants with Poor Functional Outcome (mRS 5-6) at 90±7 Days | at 90±7 days
  The secondary clinical safety outcome is the proportion of participants with poor functional outcome (severe disability or death, defined as modified Rankin Scale [mRS] score of 5-6) at 90±7 days post-treatment.
Incidence of Systemic Bleeding within 90 Days | within 90 days
  The secondary clinical safety outcome is the incidence of systemic bleeding within 90 days post-treatment, defined according to the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO) criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study can be made available to other researchers on reasonable request and after signing appropriate data sharing agreements.